CLINICAL TRIAL: NCT04883879
Title: Artificial Intelligence-based Activity Recognition and Mortality Prediction Using Circadian Rhythm, Among Cancer Patients in the Hospice Ward
Brief Title: Artificial Intelligence-based Mortality Prediction Among Cancer Patients in the Hospice Ward
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government); Taipei Medical University Hospital (Other); National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Shabbir Syed Abdul, Professor, Taipei Medical University
Other Study IDs: N201910041
Record Dates: First submitted 2021-04-28; First posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: End Stage Cancer
Keywords: Wearable Device; Actigraphy Device; Survival Prediction; Deep Learning; Artificial Intelligence; Hospice Care; Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to develop a novel deep-learning-based survival prediction model employing patient activity data recorded by a wearable device.

DETAILED DESCRIPTION:
This study aims to develop a deep-learning-based survival prediction model that utilizes patient movement data upon admission to predict their clinical outcomes: either death or discharge with stable condition. Objective data of the patients are recorded by a wearable device and documented as parameters of physical activity, angle, and spin. In addition to objective data, the investigators also document patients' Karnofsky Performance Status assessed subjectively by clinical doctors. Finally, the investigators aim to explore and describe the applicability, potential, and limitations of the survival prediction model based on patient movement data as a simple prognostic parameter in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 20 years or older admitted to the hospice care unit at Taipei Medical University Hospital
* Participants diagnosed with at least one end-stage solid tumor diseases
* Participants consented to receive hospice care

Exclusion Criteria:

* Participants aged below 20 years of age
* Participants diagnosed with leukemia or carcinoma of unknown primary
* Participants with evident signs of approaching death upon admission
* Participants with no vital signs upon admission
* Participants who continued to receive aggressive treatment despite admission to the hospice care unit

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 20 years or older who were admitted to the hospice care unit at Taipei Medical University Hospital with at least one diagnosis of end-stage solid tumor diseases.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-12-11 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Specificity and Sensitivity of using Artificial Intelligence based models for prediction of Clinical Outcomes of End-stage Cancer Patients using actigraphy data | From date of admission to hospice ward until the date of first documented discharge from hospital or date of death from any cause, whichever came first, assessed up to 1 month
  The primary outcome of the study will be to evaluate whether the analysis of the movement data captured using actigraphy device can help to predict clinical outcomes either deceased or discharged alive from hospital, with a high specificity and sensitivity, using Artificial Intelligence based prediction modelling.

CONTACTS AND LOCATIONS:
Overall Officials: Shabbir Syed-Abdul, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, TW - Taiwan, Taiwan

REFERENCES:
- [Derived] Yang TY, Kuo PY, Huang Y, Lin HW, Malwade S, Lu LS, Tsai LW, Syed-Abdul S, Sun CW, Chiou JF. Deep-Learning Approach to Predict Survival Outcomes Using Wearable Actigraphy Device Among End-Stage Cancer Patients. Front Public Health. 2021 Dec 9;9:730150. doi: 10.3389/fpubh.2021.730150. eCollection 2021. PMID 34957004